CLINICAL TRIAL: NCT01516268
Title: the Effect of Adding Sufentanyl to Bupivacaine in Transversus Abdominis Plane (TAP) Block Under the Guide of Ultrasound to Reduce the Narcotic Dosage, Side Effects and Pain in the First 24 Hours After Cesarean Delivery
Brief Title: The Effect of Adding Sufentanyl to Bupivacaine in Transversus Abdominis Plane Block to Reduce the Narcotic Dosage and Pain After Cesarean Delivery
Acronym: TAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Laleh Eslamian, Associated Prof.MD, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 886
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-02

CONDITIONS: Pain
Keywords: Cesarean Delivery; TAP block; sufentanyl; Narcotic dosages
MeSH Terms: conditions — Pain | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sufentanyl group (Active Comparator): IN case group we add 1cc sufentanyl to 20 cc bupivacain in TAP block
  Interventions: Drug: Sufentanyl
- Control group (Placebo Comparator): In control group we add 1cc salin to 20cc bupivacain in TAP block
  Interventions: Drug: Sufentanyl

INTERVENTIONS:
Drug: Sufentanyl — As intervention 1cc sufentanyl is added to bupivacain in case group for TAP block.
  As comparator 1cc normal saline is added to bupivacain in control group for Tap block.

SUMMARY:
Adding sufentanyl to bupivacain in Transversus Abdominis Plane (TAP) block under ultrasound guide can reduce narcotic dosage, side effects and pain after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* female 18 to 40 Years
* class ASA 1 and 2
* candidates for elective cesarean section

Exclusion Criteria:

* renal failure
* liver failure
* cardiac disorder
* coagulopathy
* hepatomegaly
* splenomegaly
* drug sensitivity and abuse
* morbid obesity
* smoking
* history of post operative nausea and vomiting
* motion sickness
* local hypoesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laleh Eslamian, MD, Principal Investigator — TUMS, Tehran University of Medical Sciences
Locations (1):
- Shariati hospital, TUMS, Tehran, Iran

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: Jan 2012- Dec 2013 Shariati hospital, a tertiary center
Pre-assignment Details: Exclusions were based on exclusion criteria previously mentioned.
Period: Overall Study
Arm/Group | Sufentanyl Group | Control Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 25 & 25
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanyl Group | Control Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.9 (3.4) | 29.9 (5.6) | 29.1 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Narcotic Dosage
Time Frame: 24 h
Reporting Status: Not Posted

2. Secondary Outcome: Pain
Time Frame: 24h
Reporting Status: Not Posted

3. Primary Outcome: Narcotic Dosage
Description: The total dosage of morphin consumed by the patients in sufentanil or control group.
Time Frame: over 24 hours after surgery
Measure: Mean (Standard Deviation); unit: mgm,.
Arm/Group | Sufentanyl Group | Control Group
Number analyzed (Participants) | 25 | 25
mgm,. | 37.2 (16.15) | 52.8 (16.7)

ADVERSE EVENTS:
Time Frame: 24h
Arm/Group | Sufentanyl Group | Control Group
Serious Adverse Events (participants affected / at risk) | 1/25 | 3/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanyl Group (N=25) | Control Group (N=25)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanyl Group (N=25) | Control Group (N=25)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No